CLINICAL TRIAL: NCT05167448
Title: Phase I/II Clinical Trial of ES104 in Patients With Unresectable Locally Advanced or Metastatic Colorectal Cancer Who Have Failed Systemic Therapies
Brief Title: A Study of ES104 in Patients With Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elpiscience (Suzhou) Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES104-1001
Record Dates: First submitted 2021-11-30; First posted 2021-12-22 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: ES104
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 Phase 1 (Experimental)
  Interventions: Drug: ES104
- Cohort 2 Phase 1 (Experimental)
  Interventions: Drug: ES104
- RP2D Phase 2 (Experimental)
  Interventions: Drug: ES104

INTERVENTIONS:
Drug: ES104 — ES104 is administered via Intravenous infusion, at dose of 10 mg/kg, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 2 years.
  Arms: Cohort 1 Phase 1
Drug: ES104 — ES104 is administered via Intravenous infusion, at dose of 12.5 mg/kg, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 2 years.
  Arms: Cohort 2 Phase 1
Drug: ES104 — ES104 is administered via Intravenous infusion, at dose of RP2D, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 2 years.
  Arms: RP2D Phase 2

SUMMARY:
The purpose of this open-label, Multicenter Phase I/II study is to evaluate the safety, tolerability, preliminary anti-tumor efficay, pharmacokinetics, anti-drug antibodies and biomarkers of ES104 in patients with unresectable locally advanced or metastatic colorectal cancer who have failed systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent form.
* Locally advanced or metastatic colorectal adenocarcinoma confirmed by pathology and not surgically resectable, having received systemic therapy and failed.
* At least one measurable lesion is required (RECIST v1.1)
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* Estimated life expectancy, in the judgment of the investigator, of at least 12 weeks.
* Adequate organ function, as assessed by the results of the laboratory tests specified in the protocol.
* Male and female subjects of childbearing potential must be willing to use effective contraceptive methods, from the time of signing informed consent and for the duration of study participation through 180 days following the last dose of study drug.

Exclusion Criteria:

* Receipt of any systemic antitumor therapy within 28 days prior to the first dose of study drug.
* Known history of severe allergy to any monoclonal antibody or study drug excipient.
* The subject has received or is receiving treatment in another clinical trial within 28 days prior to the first dose of study drug (except for participation in the overall survival follow-up of a study)
* Receipt of antiplatelet agents or anticoagulants for therapeutic purposes within 14 days prior to the first dose of study drug.
* Receipt of live vaccination within 28 days prior to the first dose of study drug.
* Prior history of allogeneic organ transplantation or allogeneic peripheral blood stem cell (PBSC)/bone marrow transplantation treatment.
* Subject has not recovered from all AEs of previous anticancer therapies to baseline or ≤ Grade 1 per CTCAE v5.0 before the first dose of study drug. Certain exceptions as defined in protocol apply.
* Subjects with active metastatic brain or meningeal metastases.
* Patients with other primary malignancies within 5 years before the first dose of study drug. Some exceptions as defined per protocol apply.
* Major surgery or major traumatic injury within 28 days prior to the first dose of study drug (in the judgment of the Investigator).
* History of cardiovascular disease as defined by the protocol within the past 5 years.
* History of bleeding-related illness as defined by the protocol.
* Presence of severe, unhealed or open wounds and active ulcers or untreated fractures.
* Known history of human immunodeficiency virus (HIV) virus infection and/or acquired immunodeficiency syndrome.
* Chronic active hepatitis B or active hepatitis C.
* Active infection requiring systemic therapy 14 days prior to first dose of study drug.
* Pregnant or nursing females.
* Known history of alcohol or drug abuse.
* Subjects with comorbidities or other conditions that may affect compliance with the protocol or are not suitable for participation in this study in the judgment of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: The frequency and severity of adverse events of ES104 | 1-3 years
  The safety profile of ES104 will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Phase 2: The anti-tumor activity of ES104 | 2-5 years
  The Objective Remission Rate (ORR) will be measured by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) by Investigator assessment.

SECONDARY OUTCOMES:
Phase 1: Maximum observed serum concentration (Cmax) of ES104 | 1-3 years
  Maximum observed serum concentration (Cmax) of ES104 will be measured.
Phase 1:Time to Cmax (Tmax) of ES104 | 1-3 years
  Time to Cmax (Tmax) of ES104 will be measured.
Phase 1:Area under the serum concentration time curve (AUC) of ES104 | 1-3 years
  Area under the serum concentration time curve (AUC) of ES104 will be measured.
Phase 1:The clearance of ES104 | 1-3 years
  A pharmacokinetic measurement of the volume of plasma from which ES104 is completely removed per unit time.
Phase 1: The immunogenicity of ES104 | 1-3 years
  The presence and the frequency of anti-drug antibodies (ADA) against ES104 will be measured.
Phase 1: The preliminary anti-tumor activity of ES104 | 1-3 years
  Tumor response will be measured by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) by Investigator assessment.
Phase 2: The anti-tumor activity of ES104 | 2-5 years
  Tumor response will be measured by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) by Investigator assessment.
Phase 2: The frequency and severity of adverse events of ES104 | 2-5 years
  The safety profile of ES104 will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Phase 2: The popPK profile of ES104 | 2-5 years
  The Cmin,ss、CL and Vd of ES104 will be measured.
Phase 2: The immunogenicity of ES104 | 2-5 years
  The presence and the frequency of anti-drug antibodies (ADA) against ES104 will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No